CLINICAL TRIAL: NCT04851197
Title: The Effect of Training on Testicular Cancer and Testicular Self Examination With Flipped Learning Model on Students' Knowledge and Health Beliefs
Brief Title: Flipped Learning Model on Students' Knowledge and Health Beliefs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Sevinç Taştan, Prof.Dr., Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Dogu Akdeniz Universitesi
Record Dates: First submitted 2021-04-10; First posted 2021-04-20 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Self-Examination
Keywords: Testicular Cancer; Testicular Self Examination; Flipped Learning Model; Health Beliefs; Nursing students
MeSH Terms: conditions — Self-Examination; Testicular Neoplasms

STUDY DESIGN:
Intervention Model Description: experimental study with pretest posttest control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): The students in the control group will be filled with the Introductory and Self-Testicular Examination Characteristics Question Form, "Testicular Cancer and Self Testicular Examination Knowledge Test" and "Champion's Health Belief Model Scale", which will be prepared with Microsoft teams forms before the training. Later, the students will be given an average of 20-30 minutes of training from Powerpoint presentation and video presentation. Students' questions will be answered in the last 10 minutes. After two weeks after the training, the students will be asked to fill in the "Testicular Cancer and KKTM Knowledge Test" and a Visual Analogue Scale that includes their satisfaction with the training method. After 6 weeks, "Champion's Health Belief Model Scale" will be filled out.
  Interventions: Other: Flipped Learning Model
- Intervention (Experimental): Before the training, the students in the intervention group will fill the Introductory and Characteristics Question Form on "Testicular Cancer and Self Testicular Examination Knowledge Test" and "Champion's Health Belief Model Scale". Educational materials (lecture presentation, video) will be loaded on the system in accordance with the inverted learning model, and students will be asked to come prepared for the planned lesson. Classical presentations will not be made to the students, and the education will be given in the form of question and answer discussion. After two weeks after the training, the students will be asked to fill in the "Testicular Cancer and Self Testicular Examination Knowledge Test" and a Visual Analogue Scale that includes their satisfaction with the training method. After 6 weeks, "Champion's Health Belief Model Scale" will be filled.
  Interventions: Other: Flipped Learning Model

INTERVENTIONS:
Other: Flipped Learning Model — Students in the intervention group will be given training on testicular cancer and testicular self-examination in accordance with the Flipped Learning Model. The students in the control group will receive the same training with the traditional method. It was aimed to examine the effect of the training given with the Flipped Learning Model on the students' knowledge levels and health beliefs about testicular cancer and self-testicular examination.

SUMMARY:
The aim of the training on testicular cancer and Testicular Self Examination is to increase the awareness of individuals and to develop health behaviors for early diagnosis. However, in the literature, it is seen that in the training studies conducted on this subject, mostly the training videos and presentations are made with the classical expression method. In this study, unlike other studies, the effect of the training given with the Flipped Learning Model on the knowledge and beliefs of male students regarding testicular cancer and Testicular Self Examination will be examined. It is thought that the results of the study to be obtained will guide health professionals in the selection of teaching models to increase the effectiveness of training activities to be planned for young adult males for the early diagnosis of testicular cancer.

DETAILED DESCRIPTION:
The Flipped Learning Model is a blended learning model that aims to facilitate learning with activities such as the student's pre-lesson access to educational materials such as videos and presentations through technology, and activities such as discussion, practice and problem solving during the lesson. Flipped Learning Model can be defined as a pedagological approach centered on individual learning rather than group learning. Studies show that the Flipped Learning Model has an impact on student success and satisfaction. The Flipped Learning Model has the potential to engage nursing students to meet today's needs. The complexity of students and contemporary healthcare, especially in healthcare, calls for education reform programs such as nursing highlight the students' need for problem solving, reasoning, and applying theory to practice. It manifested itself in student-based learning and case-based learning The main purpose of this study is to examine the effect of the education about testicular cancer and Testicular Self Examination given with the Flipped Learning Model on the knowledge and health beliefs of nursing students. Another aim of the study is to examine the effect of using Flipped Learning Model on student satisfaction.

The research will be carried out in Eastern Mediterranean University, Faculty of Health Sciences, Department of Nursing in the 2020-2021 academic year. Data collection will begin after the board and institution permissions are obtained for the research.

The universe of the research; Eastern Mediterranean University, Faculty of Health Sciences, Nursing Department will constitute a total of 68 male students in the 2020-2021 academic year. The sample is; After the ethics committee and institution permission is obtained, students who meet the research criteria, who are informed about the purpose of the research, and who are willing to participate in the research will be formed. The randomization of the groups to the control and intervention groups in the study will be determined by lot from the list of participants in the study.

Sample including criteria;

* Over the age of 18,
* Students who did not take the Surgical Nursing course before The data in the study were presented in the "Introductory and Self-Examination Features Questionnaire" in order to describe the characteristics of the students and testicular cancer and testicular Self Examination; It will be collected with "Testicular Cancer and Testicular Self Examination Knowledge Test" and "Champion's Health Belief Model Scale".

Research Variables Dependent variables: The dependent variables of the study were the scores obtained from the knowledge test on testicular cancer and TSE, and the Champion's Health Belief Model Scale.

Independent variables: The independent variables of the research were; Introductory features such as age, marital status, personal and family history, risk perception, information status and source of information, performing TSE, frequency of examination, and barriers to not performing TSE were created.

Data Collection Process The data of the research were collected in the fall semester of the 2020-2021 Academic Year, between December 2020 and March 2021. The data collection process was carried out in two stages, before and after the education, separately for the students in Group I and Group II. After obtaining the necessary permissions, two separate classes, Group I and Group 2, were created over Microsoft teams.

Students in Group I were asked to fill out the Introductory and Characteristics Questionnaire for TSE, the "Testicular Cancer and TSE Knowledge Test" and Champion's Health Belief Model Scale" before the training. Students were asked to come prepared to the planned lesson by uploading educational materials (lecture presentation, video) through the system in accordance with the flipped learning model. Classical presentations were not made to the students, and the education was carried out in the form of question and answer discussion, in line with the Flipped Learning Model. Two weeks after the training, the students were asked to fill in the "Testicular Cancer and TSE Knowledge Test" and the Visual Analogue Scale (VAS), which includes their satisfaction with the training method. Six weeks after the training, Champion's Health Belief Model Scale" was filled.

The students in Group II were asked to fill out the Introductory and Testicular Self-Examination Questionnaire, "Testicular Cancer and Testicular Self-Examination Knowledge Test" and Champion's Health Belief Model Scale, which were prepared with google forms before the training. Afterwards, the students were given a traditional education consisting of a Powerpoint presentation, which would last 20-30 on average. In the last 10 minutes of the lesson, the questions of the students were answered. Two weeks after the training, the students were asked to fill in the "Testicular Cancer and TSE Knowledge Test" and the Visual Analog Scale (VAS) that included their satisfaction with the training method. Six weeks after the training, the "Champion's Health Belief Model Scale" was filled.

ELIGIBILITY:
Inclusion Criteria:

Who are over the age of 18, who has not previously received testicular cancer and testicular self-examination training Being a male nursing student

Exclusion Criteria:

At any stage of the study, there is a request to withdraw from the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male nursing student who has not previously received testicular cancer and testicular self-examination training
Enrollment: 66 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Testicular Cancer and Testicular Self Examination Knowledge Test | Testicular cancer and Testicular Self Examination knowledge test will be applied baseline and two weeks after the training.
  Testicular cancer and Testicular Self Examination knowledge test was prepared by the researchers in line with the literature. In the knowledge test, there are 17 items about the incidence of testicular cancer, risk factors, symptoms, the importance of Self-Testicular Examination in early diagnosis, the frequency of performing it and how to do it. Participants will be asked to mark the questions as true, false and do not know. Expert opinion will be taken for the content validity of the prepared knowledge test. According to the results of the content validity index, the minimum and maximum points to be taken will be determined according to the number of items in the knowledge test.
Champion's Health Belief Model Scale | 6 weeks
  The Turkish reliability and validity of Champion's Health Belief Model Scale, which determines beliefs and practices for Self Testicular Examination by modifying Champion's Health Belief Model by Barnes (2000), was made by Pınar et al. (2011). The scale consists of five subscales and 26 items. Among the subscales, sensitivity: 5 items (1-5), Severity: 7 items (6-12), benefits: 3 items (13-15), barriers: 5 items (16-20) and self-efficacy: 6 items ( 21-26).

SECONDARY OUTCOMES:
Visual Analog Satisfaction Scale | 2 weeks
  Students' satisfaction with the educational method will be measured with an 11-point.Numbers between 0-10 were defined on a line, and the participants will be asked to indicate the number of satisfaction levels they feel on this line. Participants with no satisfied scored 0 and extremely satisfied participants scored 10.
  Unsatisfied participants should mark 0 points, and very satisfied participants should mark 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Sevinc Tastan, Prof. Dr., Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Health Sciences Faculty, Nursing Department, Famagusta, None Selected, Cyprus

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Le Cornet C, Lortet-Tieulent J, Forman D, Beranger R, Flechon A, Fervers B, Schuz J, Bray F. Testicular cancer incidence to rise by 25% by 2025 in Europe? Model-based predictions in 40 countries using population-based registry data. Eur J Cancer. 2014 Mar;50(4):831-9. doi: 10.1016/j.ejca.2013.11.035. Epub 2013 Dec 23. PMID 24369860
- [Background] Akar SZ, Bebis H. Evaluation of the effectiveness of testicular cancer and testicular self-examination training for patient care personnel: intervention study. Health Educ Res. 2014 Dec;29(6):966-76. doi: 10.1093/her/cyu055. Epub 2014 Sep 23. PMID 25248831
- [Background] Ugurlu Z, Akkuzu G, Karahan A, Beder A, Dogan N, Okdem S, Kav S. Testicular cancer awareness and testicular self-examination among university students. Asian Pac J Cancer Prev. 2011;12(3):695-8. PMID 21627366
- [Background] Levi F, Lucchini F, Negri E, Boyle P, La Vecchia C. Cancer mortality in Europe, 1995-1999, and an overview of trends since 1960. Int J Cancer. 2004 Jun 10;110(2):155-69. doi: 10.1002/ijc.20097. PMID 15069676
- [Background] Ugboma HA, Aburoma HL. Public awareness of testicular cancer and testicular self-examination in academic environments: a lost opportunity. Clinics (Sao Paulo). 2011;66(7):1125-8. doi: 10.1590/s1807-59322011000700001. PMID 21876962
- [Background] Betihavas V, Bridgman H, Kornhaber R, Cross M. The evidence for 'flipping out': A systematic review of the flipped classroom in nursing education. Nurse Educ Today. 2016 Mar;38:15-21. doi: 10.1016/j.nedt.2015.12.010. Epub 2015 Dec 22. PMID 26804940
- [Background] Kim HS, Kim MY, Cho MK, Jang SJ. Effectiveness of applying flipped learning to clinical nursing practicums for nursing students in Korea: A randomized controlled trial. Int J Nurs Pract. 2017 Oct;23(5). doi: 10.1111/ijn.12574. Epub 2017 Jul 25. PMID 28741796
- [Background] Hanson J. Surveying the experiences and perceptions of undergraduate nursing students of a flipped classroom approach to increase understanding of drug science and its application to clinical practice. Nurse Educ Pract. 2016 Jan;16(1):79-85. doi: 10.1016/j.nepr.2015.09.001. Epub 2015 Oct 9. PMID 26494304
- [Background] Iyigun E, Tastan S, Ayhan H, Kose G, Acikel C. Validity and reliability analysis of the planned behavior theory scale related to the testicular self-examination in a Turkish context. Postgrad Med. 2016 Jun;128(5):496-501. doi: 10.1080/00325481.2016.1182872. Epub 2016 May 10. PMID 27130481
- [Derived] Akcali K, Tastan S. The effects of flipped classroom model on knowledge, behaviour and health beliefs on testicular cancer and self-examination: a randomized controlled trial study. Health Educ Res. 2023 May 22;38(3):230-240. doi: 10.1093/her/cyad007. PMID 36843567